CLINICAL TRIAL: NCT03627104
Title: Effect of Dietary Protein and Energy Restriction in the Improvement of Insulin Resistance in Subjects With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Martha Guevara Cruz, MD and PhD., Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2373
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2018-09

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Plant Proteins, Dietary; Diet, High-Protein

STUDY DESIGN:
Intervention Model Description: The groups will receive the treatment simultaneously
Who Masked: Outcomes Assessor
Masking Description: the person who will perform the statistical analysis will be blinded from the intervention group by assigning each patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normoprotein diet with animal protein (Other): The patient will intake the diet assigned for a month
  Interventions: Dietary Supplement: Normoprotein diet with animal protein
- Normoprotein diet with vegetable protein (Other): The patient will intake the diet assigned for a month
  Interventions: Dietary Supplement: Normoprotein diet with vegetable protein
- High-protein diet with animal protein (Other): The patient will intake the diet assigned for a month
  Interventions: Dietary Supplement: High-protein diet with animal protein
- High-protein diet with vegetable protein (Other): The patient will intake the diet assigned for a month
  Interventions: Dietary Supplement: High-protein diet with vegetable protein

INTERVENTIONS:
Dietary Supplement: Normoprotein diet with animal protein — Each patient will be attended for 1 month through 4 weekly visits. Weekly menus will be delivered according to diet with percentage of standard protein (12-18%) with a predominance of animal protein (60%). Regardless of the type of protein, menus will contain the same amount of energy and concentration of carbohydrates, fats and saturated fats (less than 7%).
  Arms: Normoprotein diet with animal protein
Dietary Supplement: Normoprotein diet with vegetable protein — Each patient will be attended for 1 month through 4 weekly visits. Weekly menus will be delivered according to diet with percentage of standard protein (12-18%) with a predominance of vegetable protein (60%). Regardless of the type of protein, menus will contain the same amount of energy and concentration of carbohydrates, fats and saturated fats (less than 7%).
  Arms: Normoprotein diet with vegetable protein
Dietary Supplement: High-protein diet with animal protein — Each patient will be attended for 1 month through 4 weekly visits. Weekly menus will be delivered according to diet with high-protein percentage (25-35%) with a predominance of animal protein (60%). Regardless of the type of protein, menus will contain the same amount of energy and concentration of carbohydrates, fats and saturated fats (less than 7%).
  Arms: High-protein diet with animal protein
Dietary Supplement: High-protein diet with vegetable protein — ach patient will be attended for 1 month through 4 weekly visits. Weekly menus will be delivered according to diet with high-protein percentage (25-35%) with a predominance of vegetable protein (60%). Regardless of the type of protein, menus will contain the same amount of energy and concentration of carbohydrates, fats and saturated fats (less than 7%).
  Arms: High-protein diet with vegetable protein

SUMMARY:
The prevention of obesity and its main medical complications, such as hypertension, type 2 diabetes and cardiovascular diseases, have been become a health priority. One of the most frequent metabolic complications in obesity is the insulin resistance and is the most important risk factor for the development of coronary diseases. The weight loss induced by the restriction of dietary energy is the cornerstone of therapy for people with obesity, as it improves or even regularizes insulin sensitivity and related comorbidities. However, weight loss induced by diet also decreases lean tissue mass, which could result in adverse effects on physical function. Although, regularly recommended to increase protein intake during weight loss, there is evidence to suggest that high protein intake could have deleterious metabolic effects. On the other hand, there is an association between the type of protein consumption, mainly the concentration of branched-chain amino acids (BCAAs) and insulin resistance during the dietary energy restriction in the therapy of obesity. There are multiple factors that influence the concentration of BCAAs and insulin resistance, which can be by phenotypic or genetic modification. The phenotypic modification refers to race, sex and dietary pattern. Meanwhile, the genetic modification refers to the activity of the enzymes responsible for the catabolism of BCAAs and genetic variants, such as the polymorphisms of a single nucleotide of said enzymes. A randomized controlled trial will be conducted with 160 participants (80 women and 80 men) divided by a draw in 4 groups, each for 20 participants. A feeding plan will be assigned according to the distribution of proteins (standard or high) and type of protein (animal or vegetable). The main aim of this study is to evaluate the effect on the amount and type of dietary protein and energy restriction on insulin resistance in subjects with obesity in a period of 1 month, considering the main factors that influence the concentration of BCAAs. In this way, evidence will be provided on what type of dietary intervention is most convenient for weight loss in subjects with insulin resistance and obesity.

DETAILED DESCRIPTION:
STUDY PROGRAM The study will consist of a previous examination and 4 visits during the follow-up period.

Previous visit: pre-admission (Duration approximately 40 minutes)

1. Participants who meet the inclusion criteria will be selected. These will be captured through advertising.
2. Participants will be informed of the characteristics of the study, the risks and the benefits expected after the dietary intervention.
3. Anthropometric and body composition measurements will be made.
4. History of food frequency
5. A blood sample will be taken for the determination of glucose, insulin, total cholesterol, HDL cholesterol, LDL cholesterol, creatinine and urea nitrogen (BUN) in serum.
6. The consent letter will be signed by the participants. Subsequently according to the previous visit if insulin resistance is diagnosed according to the HOMA index (IR-HOMA), The patient will be included in the visit one of the research protocol.

Visit one:

a) Nutritional assessment (Ambulatory Patient Unit)

1. A clinical-nutritional history
2. The determination of anthropometric measurements such as weight, height and waist circumference and body composition by bioimpedance.
3. Resting energy expenditure will be determined by indirect calorimetry
4. A glucose tolerance curve will be performed for 2 hours to determine the area under the insulin and glucose curve and determination of the insulinemic and glycemic indexes.
5. A whole blood sample will be taken for the determination of the serum concentration of glucose, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, c reactive protein (CRP), insulin, leptin, and plasma amino acid profile.
6. A sample will be taken to isolate leukocytes, for the determination of the expression of enzymes related to branched-chain amino acids in leukocytes (BCAT and BCKDH).
7. The physical activity questionnaire will be carried out (IPAQ long version). The patient will be advised not to change the level of habitual physical activity
8. Patients will start consuming the diet corresponding to their group. The different menus will be delivered and explained to the patients.

7. A food guide will be given so that they have food exchange options. 8. You will be taught to fill the feed log. 9. Patients will be cited within a week.

Visit two:

1. A 24-hour dietary record.
2. Food logs will be collected and new ones will be delivered.
3. They will be given and explained the corresponding treatment menus.
4. They will be summoned in a week.

Visit three:

1. A 24-hours dietary record
2. Food logs will be collected and new ones will be delivered.
3. They will be given and explained the corresponding treatment menus.
4. They will be summoned in a week.

Visit four:

a) Nutritional assessment

1. The determination of anthropometric measurements such as weight, waist circumference and body composition measurement will be made by means of bioimpedance.
2. The resting energy expenditure will be determined by indirect calorimetry.
3. A glucose tolerance curve will be carried out for 2 hours to determine the area under the insulin and glucose curve and determination of the insulinemic and glycemic indexes.
4. A whole blood sample will be taken to determine the serum concentration of glucose, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, c-reactive protein (CRP), insulin, leptin, adiponectin and plasma amino acid profile.

6. There will be a 24-hour reminder. 7. The physical activity questionnaire will be carried out (IPAQ long version). The patient will be advised not to change the level of habitual physical activity.

8. Full feed logs will be collected. 9. It will be scheduled within fifteen days for delivery of results. Actions that will be carried out at the end of the study to maintain the continuity of the treatment

All patients after the end of the study, will be cited at 15 days where:

1. You will be given the results

ELIGIBILITY:
Inclusion Criteria:

* Adults (men and women) between the ages of 18 and 60.
* Patients with obesity (BMI ≥ 30 and ≤ 50 kg / m2) and with insulin resistance (HOMA - IR Index ≥ 2.5).
* Mexican mestizos (parents and grandparents born in Mexico).
* Patients who can read and write.

Exclusion Criteria:

* Patients with any type of diabetes.
* Patients with kidney disease diagnosed by a medical or with creatinine> 1.3 mg / dL for men and > 1.1 mg / dL for women and / or BUN> 20 mg / dL.
* Patients with acquired diseases that produce obesity and diabetes secondarily.
* Patients who have suffered a cardiovascular event.
* Patients with weight loss > 3 kg in the last 3 months.
* Patients with any catabolic diseases.
* Gravidity status
* Positive smoking
* Treatment with any medication

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Resistance insulin | Baseline to 1-month
  Change in the index HOMA-IR. The HOMA IR index will be calculated by the following equation: glucose (mg / dl) x insulin (mUI / ml) / 405 before and after of dietary intervention

SECONDARY OUTCOMES:
Amino acid profile | Baseline to 1-month
  Change in the concentration of the amino acid profile, mainly of branched chain amino acids
Change in body composition | Baseline to 1-month
  Change in fat mass, lean mass and skeletal muscle mass percentage
Change in body weight | Baseline to 1-month
  change in body weight before and after of dietary intervention
Change in waist circumference | Baseline to 1-month
  Change in waist circumference before and after of dietary intervention
Change in grip strength | Baseline to 1-month
  Change in grip strength before and after the intervention by dynamometry
Change in respiratory quotient | Baseline to 1-month
  The respiratory coefficient will be determined by indirect calorimetry
Change in glucose serum | Baseline to 1-month
  The concentration of serum glucose will be determined by autoanalyzer before and after the intervention
Change in total cholesterol serum | Baseline to 1-month
  The concentration of serum total cholesterol will be determined by autoanalyzer before and after the intervention
Change in HDL cholesterol serum | Baseline to 1-month
  The concentration of serum HDL-cholesterol will be determined by autoanalyzer before and after the intervention
Change in triglycerides serum | Baseline to 1-month
  The concentration of serum triglycerides will be determined by autoanalyzer before and after the intervention
Change in LDL cholesterol serum | Baseline to 1-month
  The concentration of serum LDL cholesterol will be determined by autoanalyzer before and after the intervention
Change in free fatty acids serum | Baseline to 1-month
  The concentration of free fatty acids will be determined before and after the intervention
Change liver function tests | Baseline to 1-month
  The concentration of serum liver enzymes will be determined by autoanalyzer before and after the intervention
Change in concentration of leptin serum | Baseline to 1-month
  The concentration of serum leptin will be determined by ELISA kit before and after the intervention
Change in concentration of adiponectin serum | Baseline to 1-month
  The concentration of serum adiponectin will be determined by ELISA kit before and after the intervention
Change in the concentration of C-reactive protein | Baseline to 1-month
  The concentration of serum C- reactive protein will be determined by autoanalyzer before and after the intervention
Change in systolic and diastolic blood pressure | Baseline to 1-month
  the blod pressure will be determined before and after the intervention
Change of the HOMA index according to the presence or absence of polymorphism related to the metabolism of branched chain amino acids (rs11548193 and rs45500792). | Baseline to 1- month
  HOMA (IR-HOMA) which is calculated glucose (mg / dl) x insulin (mUI / ml) / 405 before and after of dietary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Martha Guevara-Cruz, Dr, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Martha Guevara Cruz, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirk EP, Klein S. Pathogenesis and pathophysiology of the cardiometabolic syndrome. J Clin Hypertens (Greenwich). 2009 Dec;11(12):761-5. doi: 10.1111/j.1559-4572.2009.00054.x. PMID 20021538
- [Background] Klein S. Outcome success in obesity. Obes Res. 2001 Nov;9 Suppl 4:354S-358S. doi: 10.1038/oby.2001.142. PMID 11707565
- [Background] Wycherley TP, Moran LJ, Clifton PM, Noakes M, Brinkworth GD. Effects of energy-restricted high-protein, low-fat compared with standard-protein, low-fat diets: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2012 Dec;96(6):1281-98. doi: 10.3945/ajcn.112.044321. Epub 2012 Oct 24. PMID 23097268
- [Background] Leidy HJ, Clifton PM, Astrup A, Wycherley TP, Westerterp-Plantenga MS, Luscombe-Marsh ND, Woods SC, Mattes RD. The role of protein in weight loss and maintenance. Am J Clin Nutr. 2015 Jun;101(6):1320S-1329S. doi: 10.3945/ajcn.114.084038. Epub 2015 Apr 29. PMID 25926512
- [Background] Samson MM, Meeuwsen IB, Crowe A, Dessens JA, Duursma SA, Verhaar HJ. Relationships between physical performance measures, age, height and body weight in healthy adults. Age Ageing. 2000 May;29(3):235-42. doi: 10.1093/ageing/29.3.235. PMID 10855906
- [Background] Phillips SK, Rook KM, Siddle NC, Bruce SA, Woledge RC. Muscle weakness in women occurs at an earlier age than in men, but strength is preserved by hormone replacement therapy. Clin Sci (Lond). 1993 Jan;84(1):95-8. doi: 10.1042/cs0840095. PMID 8382141
- [Background] Brehm BJ, D'Alessio DA. Benefits of high-protein weight loss diets: enough evidence for practice? Curr Opin Endocrinol Diabetes Obes. 2008 Oct;15(5):416-21. doi: 10.1097/MED.0b013e328308dc13. PMID 18769212
- [Background] Smith GI, Yoshino J, Stromsdorfer KL, Klein SJ, Magkos F, Reeds DN, Klein S, Mittendorfer B. Protein Ingestion Induces Muscle Insulin Resistance Independent of Leucine-Mediated mTOR Activation. Diabetes. 2015 May;64(5):1555-63. doi: 10.2337/db14-1279. Epub 2014 Dec 4. PMID 25475435
- [Background] Krebs M, Krssak M, Bernroider E, Anderwald C, Brehm A, Meyerspeer M, Nowotny P, Roth E, Waldhausl W, Roden M. Mechanism of amino acid-induced skeletal muscle insulin resistance in humans. Diabetes. 2002 Mar;51(3):599-605. doi: 10.2337/diabetes.51.3.599. PMID 11872656
- [Background] Robinson MM, Soop M, Sohn TS, Morse DM, Schimke JM, Klaus KA, Nair KS. High insulin combined with essential amino acids stimulates skeletal muscle mitochondrial protein synthesis while decreasing insulin sensitivity in healthy humans. J Clin Endocrinol Metab. 2014 Dec;99(12):E2574-83. doi: 10.1210/jc.2014-2736. PMID 25222757
- [Background] Linn T, Geyer R, Prassek S, Laube H. Effect of dietary protein intake on insulin secretion and glucose metabolism in insulin-dependent diabetes mellitus. J Clin Endocrinol Metab. 1996 Nov;81(11):3938-43. doi: 10.1210/jcem.81.11.8923841.
- [Background] Sluijs I, Beulens JW, van der A DL, Spijkerman AM, Grobbee DE, van der Schouw YT. Dietary intake of total, animal, and vegetable protein and risk of type 2 diabetes in the European Prospective Investigation into Cancer and Nutrition (EPIC)-NL study. Diabetes Care. 2010 Jan;33(1):43-8. doi: 10.2337/dc09-1321. Epub 2009 Oct 13. PMID 19825820
- [Background] Tinker LF, Sarto GE, Howard BV, Huang Y, Neuhouser ML, Mossavar-Rahmani Y, Beasley JM, Margolis KL, Eaton CB, Phillips LS, Prentice RL. Biomarker-calibrated dietary energy and protein intake associations with diabetes risk among postmenopausal women from the Women's Health Initiative. Am J Clin Nutr. 2011 Dec;94(6):1600-6. doi: 10.3945/ajcn.111.018648. Epub 2011 Nov 9. PMID 22071707
- [Background] Rietman A, Schwarz J, Tome D, Kok FJ, Mensink M. High dietary protein intake, reducing or eliciting insulin resistance? Eur J Clin Nutr. 2014 Sep;68(9):973-9. doi: 10.1038/ejcn.2014.123. Epub 2014 Jul 2. PMID 24986822
- [Background] Schwingshackl L, Hoffmann G. Long-term effects of low-fat diets either low or high in protein on cardiovascular and metabolic risk factors: a systematic review and meta-analysis. Nutr J. 2013 Apr 15;12:48. doi: 10.1186/1475-2891-12-48. PMID 23587198
- [Background] Schooneman MG, Vaz FM, Houten SM, Soeters MR. Acylcarnitines: reflecting or inflicting insulin resistance? Diabetes. 2013 Jan;62(1):1-8. doi: 10.2337/db12-0466. No abstract available. PMID 23258903
- [Background] Hattersley JG, Pfeiffer AF, Roden M, Petzke KJ, Hoffmann D, Rudovich NN, Randeva HS, Vatish M, Osterhoff M, Goegebakan O, Hornemann S, Nowotny P, Machann J, Hierholzer J, von Loeffelholz C, Mohlig M, Arafat AM, Weickert MO. Modulation of amino acid metabolic signatures by supplemented isoenergetic diets differing in protein and cereal fiber content. J Clin Endocrinol Metab. 2014 Dec;99(12):E2599-609. doi: 10.1210/jc.2014-2302. PMID 25157543
- [Background] Lynch CJ, Adams SH. Branched-chain amino acids in metabolic signalling and insulin resistance. Nat Rev Endocrinol. 2014 Dec;10(12):723-36. doi: 10.1038/nrendo.2014.171. Epub 2014 Oct 7. PMID 25287287
- [Background] Serralde-Zuniga AE, Guevara-Cruz M, Tovar AR, Herrera-Hernandez MF, Noriega LG, Granados O, Torres N. Omental adipose tissue gene expression, gene variants, branched-chain amino acids, and their relationship with metabolic syndrome and insulin resistance in humans. Genes Nutr. 2014 Nov;9(6):431. doi: 10.1007/s12263-014-0431-5. Epub 2014 Sep 27. PMID 25260659
- [Derived] Gonzalez-Salazar LE, Flores-Lopez A, Serralde-Zuniga AE, Avila-Nava A, Medina-Vera I, Hernandez-Gomez KG, Guizar-Heredia R, Ontiveros EP, Infante-Sierra H, Palacios-Gonzalez B, Velazquez-Villegas LA, Ortiz-Guiterrez S, Vazquez-Manjarrez N, Aguirre-Tostado PI, Vigil-Martinez A, Torres N, Tovar AR, Guevara-Cruz M. Effect of dietary protein on serum hepcidin and iron in adults with obesity and insulin resistance: A randomized single blind clinical trial. Nutr Metab Cardiovasc Dis. 2025 May;35(5):103785. doi: 10.1016/j.numecd.2024.10.023. Epub 2024 Nov 7. PMID 39674725
- [Derived] Gonzalez-Salazar LE, Pichardo-Ontiveros E, Palacios-Gonzalez B, Vigil-Martinez A, Granados-Portillo O, Guizar-Heredia R, Flores-Lopez A, Medina-Vera I, Heredia-G-Canton PK, Hernandez-Gomez KG, Castelan-Licona G, Arteaga-Sanchez L, Serralde-Zuniga AE, Avila-Nava A, Noriega-Lopez LG, Reyes-Garcia JG, Zerrweck C, Torres N, Tovar AR, Guevara-Cruz M. Effect of the intake of dietary protein on insulin resistance in subjects with obesity: a randomized controlled clinical trial. Eur J Nutr. 2021 Aug;60(5):2435-2447. doi: 10.1007/s00394-020-02428-5. Epub 2020 Nov 3. PMID 33145643